CLINICAL TRIAL: NCT02719938
Title: Triggered Palliative Care for Advanced Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-1350; R21AG052140 (NIH); Pilot & Exploratory Project (Other: National Palliative Care Research Center)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialty Palliative Care (Experimental): Specialty inter-disciplinary Palliative Care consultation during hospitalization with post-discharge collaborative care by a Palliative Care Nurse Practitioner and outpatient primary care physician. Clinical care will be augmented by evidence-based educational materials for dementia caregivers.
  Interventions: Behavioral: Specialty Palliative Care
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Specialty Palliative Care — Specialty inter-disciplinary Palliative Care consultation during hospitalization with post-discharge collaborative care by a Palliative Care Nurse Practitioner and outpatient primary care physician. Clinical care will be augmented by evidence-based educational materials for dementia caregivers.
  Arms: Specialty Palliative Care

SUMMARY:
The objective of this study is to generate preliminary data for a large multi-site randomized clinical trial of a model of palliative care consultation for patients with advanced dementia, and for their family caregivers.

DETAILED DESCRIPTION:
Alzheimer's disease and related dementias affect 5 million Americans at an annual cost of $215 billion. Dementia is a contributing cause for 1 in 3 deaths, and is the only major cause of death with no effective prevention or treatment. Dementia-specific palliative care is needed to address the unique symptoms and treatment decisions relevant to this disease.

Investigators therefore propose to develop and pilot test a model of palliative care consultation for advanced dementia patients, triggered by hospitalization for a serious acute illness. After systematic refinement of operational protocols and tools with stakeholders, they will enroll persons with advanced dementia plus an acute illness associated with high risk of death in the coming year. Patients will be enrolled with their family decision-makers (N=60 dyads) in a randomized feasibility trial. Intervention dyads will receive specialty palliative care consultation during hospital admission, plus post-discharge collaborative care by their outpatient primary care provider and a palliative care nurse practitioner. Control dyads will receive usual care.

The research objective is to generate preliminary data for a large multi-site randomized controlled trial of a model of palliative care consultation for advanced dementia.

Specific aims are:

Aim 1: To develop a best-practice model of palliative care consultation for advanced dementia triggered by hospital admission for serious acute illness.

Aim 2: To conduct a pilot randomized trial of triggered palliative care consultation for advanced dementia (versus usual care) to demonstrate the feasibility of conducting a larger randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia from Alzheimer's or other underlying cause
* Global Deterioration Scale (GDS) Stage 5, 6 or 7
* acute illness hospitalization

Exclusion Criteria:

* No English-speaking family decision-maker
* Primary physician expects study to be too stressful for family caregiver

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hanson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing plan not written

REFERENCES:
- [Derived] Hanson LC, Kistler CE, Lavin K, Gabriel SL, Ernecoff NC, Lin FC, Sachs GA, Mitchell SL. Triggered Palliative Care for Late-Stage Dementia: A Pilot Randomized Trial. J Pain Symptom Manage. 2019 Jan;57(1):10-19. doi: 10.1016/j.jpainsymman.2018.10.494. Epub 2018 Oct 18. PMID 30342242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2016 to August 2017 enrolled dyads of hospitalized patients with late-stage dementia and family decision-makers.
Period: Overall Study
Arm/Group | Specialty Palliative Care | Control
Started | 30 | 32
Completed | 26 | 31
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Specialty Palliative Care | Control | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.0 (8.8) | 84.7 (8.7) | 83.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 10 | 17 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 21 | 23 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Hospital / Emergency Visits Per 60 Days (no. of Events/Follow-up Days)
Description: Includes emergency department visits and hospital admissions during measure interval
Time Frame: From time of hospital discharge up to 60 days
Measure: Number; unit: events per day
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
events per day | .68 | .53
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p = 0.415, t-test, 2 sided

2. Secondary Outcome: Patient Comfort End of Life in Dementia (CAD-EOLD)
Description: Comfort at the End of Life in Dementia (CAD-EOLD) instrument, consisting of 14 Likert-scaled items measuring comfort in the final phase of life with dementia. Scores range from 14-42, with higher scores indicting greater comfort.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
score on a scale | 34.8 (4.2) | 34.0 (4.1)
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p = 0.521, t-test, 2 sided

3. Secondary Outcome: Caregiver Strain
Description: Family Distress in Advanced Dementia instrument, a 21 item questionnaire designed to detect strain in family caregivers in dementia. Caregivers are asked a series of items about emotional distress, preparedness, and relations with healthcare providers scored 1-5, with higher scores indicting greater distress.
Time Frame: Interview at 60 days after hospitalization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
score on a scale | 2.3 (0.5) | 2.4 (0.5)
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p = 0.409, t-test, 2 sided

4. Secondary Outcome: Percent of Participants With Referral to Hospice or Outpatient Palliative Care From Discharge to 60 Days Follow-Up
Description: Percent of patients with referral to hospice or outpatient palliative care from discharge to 60 days follow-up from family interviews.
Time Frame: From time of hospital discharge up to 60 days
Measure: Number; unit: percentage of patients
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
percentage of patients | 25 | 3
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p = 0.019, Chi-squared

5. Secondary Outcome: Percent of Participants With Physician Orders for Life Sustaining Treatment (POLST)
Description: Percent of participants with POLST (Physician Orders for Life Sustaining Treatment) form completed and signed
Time Frame: From time of hospital discharge up to 60 days
Measure: Number; unit: percentage of participants
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
percentage of participants | 79 | 30
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Number of Palliative Care Domains in Treatment Plan
Description: Number of palliative care domains addressed in treatment plan, using the Palliative Care Domain score which is scored 0 (not addressed) or 1 (addressed) for each of 10 possible domains of a palliative care treatment plan -- prognosis, overall goals of care, physical symptoms, psychiatric symptoms, spiritual needs, and 5 treatment preferences: resuscitation, artificial feeding, intravenous fluids, antibiotics, and hospitalization. Scores are summed for a total possible score of 0-10, with higher scores indicating greater attention to palliative care needs in the treatment plan.
Time Frame: From time of hospital discharge up to 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
units on a scale | 7.6 (2.5) | 2.7 (1.7)
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Number of Participants With Burdensome Treatments
Description: Number of participants with burdensome treatments, defined as a count of participants with any use of the following treatments: feeding tube, central intravenous line, surgical procedure, intensive care transfer, ventilator use, cardiopulmonary resuscitation use at any time during the time frame of measurement.
Time Frame: From time of hospital discharge up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Specialty Palliative Care | Control
Number analyzed (Participants) | 30 | 32
Participants | 9 | 8
Statistical Analysis 1: Comparison: Specialty Palliative Care vs Control; Test type: Superiority; p = 0.516, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Specialty Palliative Care | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT02719938/Prot_SAP_000.pdf